CLINICAL TRIAL: NCT05865366
Title: Pain Trajectories and Predictors After Noncardiac Surgery in Elderly Patients: a Prospective and Observational Cohort Study
Brief Title: Pain Trajectories and Predictors After Noncardiac Surgery in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Feng Gao (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202303136
Record Dates: First submitted 2023-04-22; First posted 2023-05-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Postoperative Pain; Trajectory
Keywords: acute postoperative pain, pain trajectory, chronic pain, elderly patient
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will use group-based trajectory modeling to identify the different postoperative pain trajectory groups that exist in a mixed surgical population (non-cardiac surgery) of elderly patients during the first seven days after surgery. The aim of this study is to explore the diversity in the development of postoperative pain among elderly patients and to identify the risk factors for acute pain trajectory after surgery by investigating demographic, psychological, and clinical variables. The predictive effect of different trajectories of early postoperative acute pain on postoperative chronic pain will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for thoracic, urologic, gastrointestinal, gynecological, liver, biliary/pancreatic, or major orthopedic surgery under general anesthesia
2. Age ≥ 65 years
3. The American Society of Anaesthesiologists(ASA) I to III
4. Duration of hospitalization ≥ 72 hours

Exclusion Criteria:

1. Language disorder;
2. Hearing impairment;
3. Visual impairment;
4. The expected postoperative intubation time is more than 24 hours;
5. Critical events occurred during the perioperative period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients scheduled for thoracic, urologic, gastrointestinal, gynecological, liver, biliary/pancreatic, and major orthopedic surgeries under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Acute pain trajectories after surgery | Seven days after surgery.
  The acute pain trajectories are vectors of 7 numerical pain scores (ranging from 0 ,which indicates "no pain," to 10 , which indicates "pain as bad as you can imagine") taken over 7 days (days 1, 2, 3, 4, 5, 6, 7).
Presence of pain 3 months after surgery assessed using the Brief Pain Inventory. | 3 months after surgery
  Yes/No
Presence of pain 6 months after surgery assessed using the Brief Pain Inventory. | 6 months after surgery
  Yes/No

SECONDARY OUTCOMES:
consumption of analgesic drugs | Seven days after surgery
  the amount of analgesic drugs will be recorded
cumulative illness rating scale for geriatrics，CIR S-G | day1 before surgery
  The Cumulative Illness Rating Scale (CIRS) is utilized to assess comorbidities and comprises of 14 components, each with a severity score ranging from 0 to 4. A score of 0 indicates no damage, while a score of 1 denotes minor damage that does not impede normal activity and has a positive prognosis without treatment. A score of 2 indicates moderate damage, while a score of 3 denotes severe damage that may result in disability and necessitates immediate treatment with a poor prognosis. A score of 4 indicates fatal damage that requires urgent treatment and has a severe prognosis.
The FRAIL Scale(Fatigue, Resistance, Ambulation, Illness and Loss of Weight Index，FRAIL) | day1 before surgery
  The scale includes fatigue, resistance, ability to walk a block, concomitant illness, and weight loss. Frailty is defined by the presence of three or more of the criteria.
The douleur neuropathique 4 questionnaire(DN4) | day1 before surgery
  This questionnaire serves as a diagnostic tool for identifying neuropathic pain. It comprises 10 options, consisting of 7 self-assessment items that evaluate symptoms. The total score is 10 points, and a score of ≥ 4 indicates the possibility of neuropathic pain, while a score < 4 rules out neuropathic pain.
Mini-cog | day1 before surgery
  The Mini-Cog uses recall and clock-drawing tests to determine whether patients have cognitive impairments. A score of 0-2 indicates a positive dementia screening, while a score of 3-5 implies a negative screening, necessitating further evaluation.
The anxiety score assessed using Amsterdam preoperative anxiety and information scale | day1 before surgery
  The Amsterdam preoperative anxiety and information scale is a tool utilized to assess the level of anxiety and the amount of information patients possess before undergoing surgery.The items can be categorized into three groups - anesthesia-related anxiety score (item 1+item 2), surgery-related anxiety score (item 3+item 4), and information needs score (item 5+item 6).
  The total anxiety score is the sum of the scores for anesthesia-related anxiety and surgery-related anxiety, with higher scores indicating greater levels of anxiety.
Geriatrie depression scale，GDS-15 | day1 before surgery
  This scale serves as a diagnostic tool to screen for depression in the elderly population. A rating of 0 to 5 is within the normal range, while a score of 5 or above is indicative of a possible depression. If the total score exceeds 10, it may be appropriate to refer the individual to a psychiatric specialist for further assessment and diagnosis.
Complications within 7 days after surgery | Seven days after surgery
  Complications will be recorded.
Presence of pain before surgery assessed using the Brief Pain Inventory. | day1 before surgery
  Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China